CLINICAL TRIAL: NCT02700997
Title: Uterosacral Ligament Suspension: A Radiographic Study of Anatomy and Suture Location
Brief Title: Uterosacral Ligament Suspension Clip
Acronym: USLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-092
Record Dates: First submitted 2016-01-06; First posted 2016-03-07 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vascular clip (Experimental): Application of a clip to dissolvable sutures.
  Interventions: Device: Vascular Clip

INTERVENTIONS:
Device: Vascular Clip — Application of a titanium vascular clip (size small) to the base of each delayed absorbable suture placed at the vaginal apex on the internal vaginal side to help in identification by imaging
  Other Names: Clip

SUMMARY:
This study seeks to gain a more thorough understanding of the postoperative location of the sutures placed during uterosacral ligament suspension. Characterization of the surrounding anatomy in a living model will enhance surgical technique by delineating safer suture locations and decrease the incidence of morbid complications for patients.

DETAILED DESCRIPTION:
Uterosacral ligament suspension Is a commonly performed procedure to support the vaginal apex at the time of pelvic reconstructive surgery for pelvic organ prolapse (POP). Despite being a well established durable option for patients, there is little research detailing ligament suspension suture location in the living model. The available literature is limited to cadaveric studies, which suggest suture placement is in close proximity to vital structures such as the ureter, blood vessels, rectum and nerves.

This study seeks to describe suture location in relation to the surrounding anatomy in postoperative patients following high uterosacral ligament suspension. The secondary aim is to determine safe zones for suture placement.

Seventeen women (aged 18-85) under the care of Cincinnati Urogynecology Associates, a physician group of TriHealth, who have chosen vaginal hysterectomy with uterosacral ligament suspension (USLS) as the treatment choice for pelvic organ prolapse (POP) will be enrolled.

At the time of surgery, a titanium vascular clip (size small) will be applied to the base of each delayed absorbable suture placed at the vaginal apex on the internal vaginal side to help in identification by imaging.

On postoperative day (POD) 1, patients will undergo CT pelvis scans. The CT scan will involve administration of IV contrast for imaging of the ureters and vascular structures. The clip will fall off when the sutures dissolve at 12 weeks postoperatively. All patients will be asked to complete a lower extremity neurological questionnaire preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-85 with pelvic organ prolapse (POP) who have elected uterosacral ligament suspension (USLS) for treatment

Exclusion Criteria:

* contraindication to computed tomography (CT), or intravenous (IV) contrast
* those with claustrophobia
* previous POP surgery
* previous pelvic surgery to the fallopian tubes, ovaries, or rectum
* previous pelvic radiation
* known pelvic inflammatory disease or endometriosis
* those with preexisting ureteral or vascular pathology or sacral anatomic abnormality
* those with connective tissue disorders
* those with preexisting neuropathy, chronic lower extremity pain disorders, or neurological disorders
* those with renal anomalies such as pelvic kidney, duplication of the collecting system, prior nephrectomy
* those with allergy to titanium
* removal of the uterosacral sutures due to ureteral obstruction intraoperatively

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith BC, Herfel CV, Yeung J, Shatkin-Margolis A, Crisp CC, Kleeman SD, Pauls RN. Uterosacral Ligament Suspension: A Radiographic Study of Suture Location in Live Subjects. Female Pelvic Med Reconstr Surg. 2020 Sep;26(9):541-545. doi: 10.1097/SPV.0000000000000629. PMID 30180050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vascular Clip
Started | 17
Completed | 15
Not Completed | 2
Not completed — Did not undergo CT imaging | 1
Not completed — No CT measurement - pelvic calcification | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vascular Clip
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
BMI [Median (Full Range); unit: kg/m^2] | 28 [21.8 to 43.9]

OUTCOME MEASURES:

1. Primary Outcome: Suture Location in Relation to the Surrounding Anatomy
Description: Measurement between internal iliac complex and proximal suture; measurement between ureter and proximal/distal suture.
Time Frame: 1 day after surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Vascular Clip
Number analyzed (Participants) | 15
cm
  Internal iliac complex from right proximal suture | 2.5 (0.5)
  Internal iliac complex from left proximal suture | 2.8 (0.7)
  Right ureter from right proximal suture | 2.2 (0.5)
  Right ureter from right distal suture | 2.2 (0.4)
  Left ureter from left proximal suture | 2.4 (0.6)
  Left ureter from left distal suture | 2.5 (0.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Vascular Clip
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT02700997/Prot_SAP_000.pdf